CLINICAL TRIAL: NCT07015931
Title: Efficacy of 0.025% Retinoic Acid Cream Compared to 0.1% Adapalene Cream on Mild Acne Vulgaris, as Well as Safety Profile and Post-Acne Sequelae in Fitzpatrick Skin Types III-V: A Randomized Double-Blind Clinical Trial Using the Split-Face Method
Brief Title: Efficacy, Safety Profile, and Post-Acne Sequelae of 0.025% Retinoic Acid Cream vs. 0.1% Adapalene Cream in Mild Acne Vulgaris in Fitzpatrick Skin Types III-V
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Reisa Reshinta, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-08-1369
Record Dates: First submitted 2025-05-26; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; mild acne; retinoic acid 0.025%; adapalene 0.1%; topical retinoids; acne treatment; Fitzpatrick skin type III-V; post inflammatory hyperpigmentation; post acne erythema; post acne scarring; adverse effects of retinoids; clinician erythema assessment; randomized controlled trial; acne lesion count; acne sequelae
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with 0.025% Retinoic Acid Cream (Split-Face Design) (Experimental): Participants will apply 0.025% retinoic acid cream half finger tip unit on one randomized side of the face every night for 12 weeks.
  Interventions: Drug: retinoic acid cream 0.025%
- Treatment with 0.1% Adapalene Cream (Split-Face Design) (Experimental): Participants will apply 0.1% adapalene cream half finger tip unit on one randomized side of the face every night for 12 weeks.
  Interventions: Drug: adapalene cream 0.1%

INTERVENTIONS:
Drug: retinoic acid cream 0.025% — half finger tip unit
  Arms: Treatment with 0.025% Retinoic Acid Cream (Split-Face Design)
Drug: adapalene cream 0.1% — half finger tip unit
  Arms: Treatment with 0.1% Adapalene Cream (Split-Face Design)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness, safety profile, and post-acne sequelae of 0.025% retinoic acid cream versus 0.1% adapalene cream for mild acne vulgaris in individuals with Fitzpatrick skin types III-V.

Main research questions are:

1. How does 0.025% retinoic acid cream compare to 0.1% adapalene cream in reducing the total number of acne lesions in patients with mild acne vulgaris and Fitzpatrick skin types III-V?
2. What is the severity of adverse effects that occur on the facial side treated with 0.1% adapalene cream and the facial side treated with 0.025% retinoic acid cream in patients with mild acne vulgaris and Fitzpatrick skin types III-V?
3. What is the severity of post-inflammatory hyperpigmentation (PIH) that occurs on the facial side treated with 0.1% adapalene cream and the facial side treated with 0.025% retinoic acid cream in patients with mild acne vulgaris and Fitzpatrick skin types III-V?
4. What is the severity of post-acne erythema (PAE) that occurs on the facial side treated with 0.1% adapalene cream and the facial side treated with 0.025% retinoic acid cream in patients with mild acne vulgaris and Fitzpatrick skin types III-V?
5. What is the quantity, type, and severity of post-acne scarring (PAS) that occurs on the facial side treated with 0.1% adapalene cream and the facial side treated with 0.025% retinoic acid cream in patients with mild acne vulgaris and Fitzpatrick skin types III-V?

Participants will:

* Undergo baseline assessments, including acne lesion count, hyperpigmentation index, Clinician Erythema Assessment (CEA) scale, and post-acne scarring grading on each facial side.
* Apply 0.025% retinoic acid cream and 0.1% adapalene cream on different facial sides as per randomization, every night for 12 weeks.
* Record daily adverse effects per facial side, lesion manipulation frequency, and sun exposure duration
* Attend follow-up visits every 4 weeks for acne lesion count, hyperpigmentation index, CEA scale, post-acne scarring grading, and assessment of adverse effect severity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild acne vulgaris, defined as fewer than 20 comedonal lesions, fewer than 15 inflammatory lesions, or a total lesion count of 30 or less, with a difference in total lesion count between the two sides of the face ≤ 5 lesions.
* Minimum age of 15 years.
* Indonesian individuals with Fitzpatrick skin types III-V.
* Willing to participate in the study by signing an informed consent form.

Exclusion Criteria:

* History of routine application of topical agents containing active ingredients on the face within the past 2 weeks.
* History of oral antibiotic use within the past 2 weeks.
* History of systemic retinoid use within the past 3 months.
* Currently pregnant or breastfeeding.
* Using oral contraceptives at the time of assessment.
* Presence of other dermatologic conditions on the face aside from acne vulgaris.
* Having sensitive facial skin classified as rosacea-type, stinging-type, or allergic-type.
* Unwilling to discontinue topical active agent therapy that has been used routinely for at least 2 weeks prior to study participation.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage reduction in total acne lesions between the 0.025% tretinoin cream group and the 0.1% adapalene cream group | from enrollment to the end of treatment at 12 weeks
  The percentage reduction was calculated by comparing the total number of lesions at 12 weeks to baseline counts

SECONDARY OUTCOMES:
Severity profile of adverse effects | from enrollment to the end of treatment at 12 weeks
  Mild: presence of subjective symptoms such as itching or burning sensation without any objective signs (e.g., erythema or desquamation);
  Moderate: presence of both subjective symptoms and objective signs, but not interfering with daily activities or treatment adherence;
  Severe: presence of subjective and objective signs that are bothersome and interfere with the patient's comfort or treatment adherence
  The proportion for each severity grade will be presented as a percentage.
Hyperpigmentation index profile | from enrollment to the end of treatment at 12 weeks
  The hyperpigmentation index was calculated by multiplying the intensity score of each lesion-assessed using the Taylor Hyperpigmentation Scale-by the total number of lesions. The final index was obtained by averaging the results across all affected sites. The minimum possible score is 0, and the maximum score is 9. A higher score indicates more severe post-acne hyperpigmentation experienced by the study subjects.
Post acne erythema profile | from enrollment to the end of treatment at 12 weeks
  Post-acne erythema was assessed using the Clinician Erythema Assessment (CEA) scale, which grades erythema severity into five categories: clear, almost clear, mild, moderate, and severe. The proportion for each severity grade will be presented as a percentage.
Profile of post-acne scar type | from enrollment to the end of treatment at 12 weeks
  The types of post-acne scars recorded included icepick, rolling, boxcar, hypertrophic, keloid, and papular scars. The proportion of each scar type was calculated and will be presented as percentage.
Severity profile of post acne scarring | from enrollment to the end of treatment at 12 weeks
  Additionally, the severity of post-acne scarring was graded as macular, mild, moderate, or severe based on clinical evaluation. The proportion for each grade will be presented as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, DKI Jakarta, Indonesia